CLINICAL TRIAL: NCT04618627
Title: Role of Lung Ultrasonography in Prediction of the Seveity and the Need for Surfactant Administration in Neonates With Respiratory Distress Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Elyan Ahmed, doctor, Assiut University
Other Study IDs: RLUSIRDS
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Lung Ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: lung ultrasound — Role of lung ultrasonography in prediction of the seveity and the need for surfactant administration in neonates with respiratory distress syndrome.

SUMMARY:
We aim to identify the diagnostic role of a lung ultrasonography (LUS) score to predict the severity and the need for surfactant therapy in newborns with respiratory distress syndrome (RDS), and to compare it with a chest X-ray score.

DETAILED DESCRIPTION:
Respiratory distress syndrome (RDS) is a common problem in preterm infants. This condition is caused by deficiency of pulmonary surfactant in an immature lung and is related to morbidity and mortality in preterm infants. The incidence of RDS increases with the decreasing of gestational age (GA). The National Institute of Child Health and Human Development Neonatal Research Network reports a 93 percent incidence of RDS in a cohort of extremely preterm infants (GA 28 weeks or below)1. Although the risk is lower, RDS occurs even in a significant number of late preterm infants2. Diagnosis of RDS is based on clinical manifestations, arterial blood gas and chest X-ray findings. Chest X-ray is considered a first-line imaging test for diagnosis of RDS2. Chest X-ray findings, however, are not related to the respiratory prognosis3 .

Recently, lung ultrasonography (LUS) has been used in critically ill patient and it has become an important tool for neonatologists4. Specific LUS patterns have been described for typical neonatal respiratory conditions such as RDS5, transient tachypnea of the newborn (TTN)6, meconium aspiration syndrome (MAS)7, and pneumothorax8,9.As reported in The Consensus Conference on lung ultrasound, both LUS and chest X-ray are accurate in the diagnosis of RDS and TTN in neonates10.

Surfactant replacement therapy is crucial in the management of RDS. Recent guidelines recommend to treat affected babies with early nasal continuous positive airway pressure (nCPAP) and early selective surfactant administration10. The European Association of Perinatal Medicine and the American Academy of Pediatrics advise surfactant administration when oxygen requirement increases despite early nCPAP treatment11,12. Some studies have recently highlighted the usefulness of LUS in predicting neonatal intensive care unit admission or the need for mechanical ventilation13,14 or nCPAP failure15. Many scores based on LUS findings have proved their reliability in adult critical care16,17. In the neonatal field few studies presented chest X-ray derived scores18 or directly compared LUS with chest ray. There are no data, to our knowledge, that compare the accuracy of LUS with chest X-ray in predicting the need for surfactant administration in infants with RDS18-20.

Basically, each lung was divided into 3 areas (upper anterior, lower anterior, and lateral) and examined using a linear microprobe through both transverse and longitudinal scans. For each lung area, a 0- to 3-point score was given (total score ranging from 0-18). The LUS score encompassed signs typical of TTN and RDS21-22 . and described the total spectrum of possible conditions (a normal aerated lung, an interstitial pattern, an alveolar pattern, and consolidation). In details, the LUS score was assigned as follows:0 indicates A-pattern (defined by the presence of the only A-lines); 1, B-pattern (defined as the presence of ≥3 well-spaced B-lines); 2, severe B pattern (defined as the presence of crowded and coalescent B lines with or without consolidations limited to the subpleural space); and 3, extended consolidations. A-lines represent reflection of pleura due to ultrasound diffusing through an airfilled lung; B-lines are due to fluid filling the interstitium (and the alveolar space if they become confluent)23,24.

ELIGIBILITY:
Inclusion Criteria:

* • Gestational age < 28 weeks.

  * Birth weight <1000 grams.
  * Newborns diagnosed only with RDS clinically and by chest X-Ray findings

Exclusion Criteria:

* • Gestational age ≤ 28 weeks.

  * Birth weight ≤ 1000 grams.
  * Newborns with congenital anomalies.

Ages: 1 Hour to 1 Month | Sex: All
Age Groups: Child
Study Population: Gestational age < 28 weeks.
  * Birth weight <1000 grams.
  * Newborns diagnosed only with RDS clinically and by chest X-Ray findings
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity lung ultrasound examination in identifying the severity and need for surfactant administration in neonates with RDS | baseline
  Sensitivity and specificity lung ultrasound examination in identifying the severity and need for surfactant administration in neonates with RDS

SECONDARY OUTCOMES:
Compare point-of-care lung ultrasound with chest x ray in the rate of detection of RDS in neonates. | baseline
  Compare point-of-care lung ultrasound with chest x ray in the rate of detection of RDS in neonates.

CONTACTS AND LOCATIONS:
Overall Officials: fatma ali, professor, Study Director — assiut university children hospital

REFERENCES:
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Kurl S, Heinonen KM, Kiekara O. The first chest radiograph in neonates exhibiting respiratory distress at birth. Clin Pediatr (Phila). 1997 May;36(5):285-9. doi: 10.1177/000992289703600506. PMID 9152555
- [Background] Copetti R, Cattarossi L, Macagno F, Violino M, Furlan R. Lung ultrasound in respiratory distress syndrome: a useful tool for early diagnosis. Neonatology. 2008;94(1):52-9. doi: 10.1159/000113059. Epub 2008 Jan 15. PMID 18196931
- [Background] Copetti R, Cattarossi L. The 'double lung point': an ultrasound sign diagnostic of transient tachypnea of the newborn. Neonatology. 2007;91(3):203-9. doi: 10.1159/000097454. Epub 2006 Dec 6. PMID 17377407
- [Background] Piastra M, Yousef N, Brat R, Manzoni P, Mokhtari M, De Luca D. Lung ultrasound findings in meconium aspiration syndrome. Early Hum Dev. 2014 Sep;90 Suppl 2:S41-3. doi: 10.1016/S0378-3782(14)50011-4. PMID 25220126
- [Background] Migliaro F, Sodano A, Capasso L, Raimondi F. Lung ultrasound-guided emergency pneumothorax needle aspiration in a very preterm infant. BMJ Case Rep. 2014 Dec 14;2014:bcr2014206803. doi: 10.1136/bcr-2014-206803. PMID 25512394
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031